CLINICAL TRIAL: NCT05855213
Title: RolE of High Velocity Nasal Insufflation in imrpoVing wEaning Success in Respiratory Failure Patients (REVIVER)
Brief Title: HVNI for Successful Weaning in Respiratory Failure
Acronym: REVIVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Salama Sadaka, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010594
Record Dates: First submitted 2023-04-08; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Failure; Weaning Failure
Keywords: HVNI; non-invasive ventilation; weaning failure; extubation; respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: This is a single center prospective randomized controlled open label trial of high velocity nasal insufflation (HVNI) in the immediate post-extubation period versus noninvasive positive pressure ventilation (NIPPV). Allocation arm failure , assessed after 72 hours of extubation, will be the primary outcome. Cross-over from HVNI to NIPPV may be allowed in case of HVNI failure and potential benefit as judged by the treating clinical team prior to reintubation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Velocity Nasal Insufflation (HVNI) (Experimental): HVNI (Precision Flow; Vapotherm®, Inc, Exeter, NH) will be delivered using a small-bore nasal cannula initiated at a flow rate set to 35 L/min, temperature of 35-37°C and FiO2 at 1.0. Adjustments in flow (up to 40 L/min) and temperature will be titrated to optimize patient's comfort.
  The target parameters after initiation will be as follows:
  1. RR< 25 bpm
  2. HR< 120 bpm
  3. SpO2 92-94%
  Interventions: Device: High Velocity Nasal Insufflation
- Non-invasive positive pressure ventilation (NIPPV) (Active Comparator): NIPPV will be initiated with an oronasal mask, with inspiratory and expiratory positive airway pressures (IPAP, EPAP) set at IPAP 10-20 cm H2O and EPAP 5-7 cm H2O to be titrated according to patient's response and comfort. FiO2 will be initiated at 1.0 for noninvasive positive-pressure ventilation.
  The target parameters after initiation will be as follows:
  1. RR< 25 bpm
  2. HR< 120 bpm
  3. SpO2 92-94%
  Interventions: Device: Non-invasive positive pressure ventilation

INTERVENTIONS:
Device: High Velocity Nasal Insufflation — A relatively new respiratory support modality which delivers very high velocity flows. This improves ventilatory efficiency via washing out carbon dioxide occupying the anatomical dead space of the upper airways.
  Other Names: HVNI
  Arms: High Velocity Nasal Insufflation (HVNI)
Device: Non-invasive positive pressure ventilation — An established non-invasive ventilation method via delivery of an expiratory positive airway pressure and inspiratory positive airway pressure.
  Other Names: NIPPV
  Arms: Non-invasive positive pressure ventilation (NIPPV)

SUMMARY:
The goal of this randomized active-controlled study is to investigate the role of high velocity nasal insufflation (HVNI) in the immediate post-extubation period and compare it with non-invasive positive pressure ventilation (NIPPV) as regards to weaning success rate. The study will recruit those who have been on invasive mechanical ventilation for at least 3 days and with a high risk of weaning failure.

DETAILED DESCRIPTION:
This is a single center prospective randomized controlled open label trial of high velocity nasal insufflation (HVNI) in the immediate post-extubation period versus noninvasive positive pressure ventilation (NIPPV). After at least 72 hours from intubation, for respiratoy failure, those who are considered to be eligible for weaning from mechanical ventilation based on the weaning protocol but are at high risk for extubation failure will be randomized to either HVNI or NIPPV. Data on the respiratory and cardiovascular status will be continuously monitored and recorded thereafter.

The primary outcome measure will be failure of either arm within 72 hours of initiation, leading to reintubation (or crossover only from a failed HVNI allocation to NIV based on clinical judgement to avoid reintubation in selected cases). Secondary outcomes to be investigated include: 1) Failure of HVNI or NIPPV after 72 hours from initiation, 2) hospital mortality, 3) length of ICU stay, 4) length of hospital stay, 5) incidence of ventilator associated pneumonia, 6) patient tolerance and comfort, and 7) ICU readmission or mortality at 28-days post hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

High risk of extubation failure (one or more of the following):

1. Age >65 years old
2. BMI >30
3. APACHE II score at extubation >12
4. ≥2 comorbidities
5. Endotracheal intubation > 7 days
6. ≥1 failed attempts at disconnection from mechanical ventilation
7. Chronic lung disease e.g., COPD, OHS, etc.
8. Underlying left ventricular dysfunction
9. Non-minimal airway secretions

Exclusion Criteria:

1. Non-respiratory failure patients
2. Patients judged to need a tracheostomy (poor airway reflexes or copious secretions)
3. Patients who cannot tolerate an oral or nasal interface (facial trauma or perforated nasal septum)
4. Patients with increased risk of aspiration, agitation, or uncooperativeness
5. End stage disease with life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Failure of HVNI / NIPPV within 72 hours of initiation | within 72 hours from start of either allocated modality
  need to withdraw allocated respiratory support modality based on predefined arm failure criteria

SECONDARY OUTCOMES:
Failure of HVNI / NIPPV after 72 hours of initiation | beyond 72 hours from start of either allocated modality
  need to withdraw allocated respiratory support modality based on predefined arm failure criteria
Length of ICU stay | Through study completion, an average of 1 year
  number of days from ICU admission to discharge
Length of Hospital stay | Through study completion, an average of 1 year
  number of days from hospital admission to discharge
Hospital Mortality | Through study completion, an average of 1 year
  mortality rate in each allocated arm
Patient tolerance and comfort | within 72 hours from start of either allocated modality
  Rate of tolerance to allocated respiratoy support modality in each arm
Incidence of ventilator associated pneumonia (VAP) | beyond 48 hours from start of invasive mechanical ventilation
  percentage of participants developing VAP
ICU readmission or mortality post hospital discharge | 28 days after hospital discharge
  percentage of participants from each arm needing ICU readmission or dying within 4 weeks of hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Diseases Department, Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Upon reasonable request